CLINICAL TRIAL: NCT01787409
Title: Effect of Vitamin D Replacement on Tumor Response and Survival Parameters for Vitamin D Insufficient Patients With Cancer
Brief Title: Cholecalciferol in Improving Survival in Patients With Newly Diagnosed Cancer With Vitamin D Insufficiency
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LS1293; NCI-2013-00037 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); LS1293 (Other: Mayo Clinic); P50CA097274 (NIH); 12-007862 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Aggressive Non-Hodgkin Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-Cell Lymphoma; Chronic Lymphocytic Leukemia; Diffuse Large B-Cell Lymphoma; Enteropathy-Associated T-Cell Lymphoma; Hepatosplenic T-Cell Lymphoma; Mature T-Cell and NK-Cell Non-Hodgkin Lymphoma; Mediastinal (Thymic) Large B-Cell Lymphoma; Nasal Type Extranodal NK/T-Cell Lymphoma; Peripheral T-Cell Lymphoma, Not Otherwise Specified; Primary Cutaneous Anaplastic Large Cell Lymphoma; Refractory Anaplastic Large Cell Lymphoma; Small Lymphocytic Lymphoma; Subcutaneous Panniculitis-Like T-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Enteropathy-Associated T-Cell Lymphoma; Lymphoma, T-Cell; Lymphoma, Extranodal NK-T-Cell; Lymphoma, Primary Cutaneous Anaplastic Large Cell; Subcutaneous panniculitis-like T-cell lymphoma | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (cholecalciferol) (Experimental): Vitamin D sufficient patients receive no intervention. Vitamin D insufficient patients receive cholecalciferol PO once weekly for 12 weeks and then once monthly for a total of 36 months.
  Interventions: Dietary Supplement: Cholecalciferol; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Dietary Supplement: Cholecalciferol — Given PO
  Other Names: 9,10-Secocholesta-5,7,10(19)-trien-3-ol; Calciol; Delsterol; Vitamin D3
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This partially randomized clinical trial studies cholecalciferol in improving survival in patients with newly diagnosed cancer with vitamin D insufficiency. Vitamin D replacement may improve tumor response and survival and delay time to treatment in patients with cancer who are vitamin D insufficient.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if vitamin D replacement in vitamin D insufficient patients with newly diagnosed untreated diffuse large B-cell lymphoma (DLBCL) can improve event free survival at 12 months to be equivalent to that of a control population of vitamin D sufficient patients. (Study I) II. To assess the percentage of patients requiring treatment with conventional therapy at 36 in months in vitamin D insufficient patients with early stage chronic lymphocytic leukemia (CLL) being managed with observation who undergo vitamin D replacement. (Study II)

SECONDARY OBJECTIVES:

I. To assess the effect of vitamin D replacement in vitamin D insufficient patients with newly diagnosed untreated DLBCL on overall survival. (Study I) II. To assess the effect of vitamin D replacement in vitamin D insufficient patients with newly diagnosed untreated DLBCL on event free survival. (Study I) III. To assess the effect of vitamin D replacement in vitamin D insufficient patients with newly diagnosed untreated T cell lymphoma on event free and overall survival. (Study I) IV. To assess the effect of vitamin D replacement in vitamin D insufficient CLL patients on Bio-r response rate and overall response rate. (Study II) V. To assess time to treatment and overall survival in vitamin D insufficient CLL patients who received vitamin D replacement. (Study II)

TERTIARY OBJECTIVES:

I. To study immune effector cells (lymphocytes, monocytes), serum cytokines, and tumor cells from vitamin D deficient and sufficient patients to learn the effects of vitamin D on both tumor cells and the patient's immune system. (Study I-II)

OUTLINE:

Vitamin D sufficient patients receive no intervention. Vitamin D insufficient patients receive cholecalciferol orally (PO) once weekly for 12 weeks and then once monthly for a total of 36 months.

After completion of study treatment, patients are followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed aggressive lymphoma or CLL/small lymphocytic lymphoma (SLL) that meets disease specific criteria below:
* Study 1 - Aggressive lymphoma

  * Newly diagnosed de-novo DLBCL or primary mediastinal B-cell lymphoma that will be treated with an anthracycline-containing regimen (rituximab-cyclophosphamide, doxorubicin hydrochloride, prednisone [R-CHOP] or equivalent); patients with composite lymphomas can also be enrolled as long as they have large cell component and will be treated with an anthracycline; in addition, patients with "B cell lymphoma, unclassifiable, with features intermediate between diffuse large B cell lymphoma and Burkitt lymphoma" or post-transplant DLBCL are also eligible as long as they meet other criteria; patients with typical Burkitt lymphoma are not eligible

    * NOTE: patients can be enrolled up through day 1 of cycle 3 of therapy; the patient is permitted to participate in any other therapeutic therapy for their disease as long as it does not concern vitamin D; patients can begin their chemotherapy while awaiting vitamin D results and treatment arm assignment or
  * Newly diagnosed untreated peripheral T-cell non-Hodgkin lymphoma (NHL) that will be treated with chemotherapy; NOTE: patients can be enrolled up through day 1 of cycle 3 of therapy; this includes the following disease types:

    * Peripheral T cell lymphoma, unspecified
    * Anaplastic large cell lymphoma (T and null cell type)
    * Extranodal NK/T-cell lymphoma, nasal type
    * Enteropathy-type T-cell lymphoma
    * Hepatosplenic T-cell lymphoma
    * Subcutaneous panniculitis-like T-cell lymphoma
    * Angioimmunoblastic T-cell lymphoma
    * Anaplastic large cell lymphoma - primary cutaneous type and
  * Willing to provide tissue for correlative research purposes
* Study 2 - CLL/SLL

  * Newly diagnosed (< 12 months from pre-registration on this study) CLL according to the National Cancer Institute (NCI) criteria or SLL according to the World Health Organization (WHO) criteria; this includes previous documentation of:

    * Biopsy-proven small lymphocytic lymphoma
    * Diagnosis of CLL according to NCI working group criteria as evidenced by all of the following:

      * Peripheral blood lymphocyte count of > 5,000/mm^3; if present, prolymphocytes should be < 55%
      * Immunophenotyping consistent with CLL defined as:

        * The predominant population of lymphocytes share both B-cell antigens (cluster of differentiation [CD]19, CD20, or CD23) as well as CD5 in the absence of other pan-T-cell markers (CD3, CD2, etc.)
        * Dim surface immunoglobulin expression
        * Restricted surface kappa or lambda light chain expression
      * Before diagnosing CLL or SLL, mantle cell lymphoma must be excluded by demonstrating a negative fluorescent in situ hybridization (FISH) analysis for t(11;14)(immunoglobulin H [IgH]/cyclin D 1 [CCND1]) on peripheral blood or tissue biopsy or negative immunohistochemical stains for cyclin D1 on involved tissue biopsy
  * Rai stage 0 or 1
  * Previously untreated
  * Asymptomatic with the plan for observation
  * Life expectancy of at least 24 months
  * Willing to provide tissue for correlative research purposes
* Both Studies:
* Capable of swallowing intact study medication capsules
* Serum calcium < 11 mg/dL; note: patients with hypercalcemia can be enrolled after the calcium is corrected with standard of care treatments
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)

  * Note: During the Active Monitoring Phase of a study (i.e., active treatment and observation), participants must be willing to return to the consenting institution for follow-up
* Willing to provide blood samples for correlative research purposes
* Vitamin D level (25 hydroxy D2 + hydroxyl D3) confirmed by central laboratory review

Exclusion Criteria:

* Patients with Burkitt lymphoma or any patient receiving rituximab-cyclophosphamide, vincristine, doxorubicin, high-dose methotrexate / ifosfamide, etoposide, high-dose cytarabine (R- CODOXM/IVAC)
* Patients who previously had indolent lymphoma and now at a separate episode have large cell NHL (i.e. transformation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 565 (Actual)
Dates: Start 2013-03-06 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Event free survival (EFS) (Study I) | Time from study registration to lymphoma progression, initiation of new anti-lymphoma therapy after completion or cessation of the original anthracycline based treatment, or death due to any cause, assessed at 12 months
  The proportion of successes will be estimated separately in the groups by the number of successes divided by the total number of evaluable patients. 95% confidence intervals for the true success proportion will be calculated by the exact binomial method.
Treatment free status (Study II) | At 36 months
  The proportion of successes will be estimated separately in the groups by the number of successes divided by the total number of evaluable patients. 95% confidence intervals for the true success proportion will be calculated by the exact binomial method.

SECONDARY OUTCOMES:
Bio-R response rate (Study II) | Up to 5 years
  Bio-R response rate will be calculated as the number of patients with Bio-R response divided by the number of evaluable patients. If a sufficient number of Bio-R responses are seen, differences in Bio-R rate between the two study groups will be evaluated using Fisher's exact test.
EFS time (Study I) | From study registration to lymphoma progression, initiation of new anti-lymphoma therapy after completion or cessation of the original anthracycline based treatment, or death due to any cause, assessed up to 5 years
  The distribution of event-free survival time in each group will be estimated using the method of Kaplan-Meier. Differences between the groups will be evaluated using Cox proportional hazard models.
OS (Study II) | From registration to death due to any cause, assessed up to 5 years
  The distribution of survival time will be estimated using the method of Kaplan-Meier. Differences between the groups will be evaluated using Cox proportional hazard models. These models will be assessed both unadjusted and adjusted for Rai stage and FISH [favorable (13q-, +12, no abnormalities) vs. unfavorable (11q-, 17p-)].
Overall response rate (Study II) | Up to 5 years
  Exact binomial 95% confidence intervals for the true overall response rate will be calculated. If a sufficient number of responses are seen, differences in overall response rate between the two study groups will be evaluated using Fisher's exact test.
Overall survival (OS) time (Study I) | From registration to death due to any cause, assessed up to 5 years
  The distribution of survival time will be estimated using the method of Kaplan-Meier. Differences between the groups will be evaluated using Cox proportional hazard models. These models will be assessed both unadjusted and adjusted for Rai stage and FISH [favorable (13q-, +12, no abnormalities) vs. unfavorable (11q-, 17p-)].
Time to first treatment (Study II) | From study registration to initiation of anti-CLL therapy, assessed up to 5 years
  The distribution of time to first treatment will be estimated using the method of Kaplan-Meier. Differences between the two study groups will be evaluated using Cox proportional hazard models. These models will be assessed both unadjusted and adjusted for Rai stage and FISH [favorable (13q-, +12, no abnormalities) vs. unfavorable (11q-, 17p-)].

OTHER OUTCOMES:
Gene expression profiles | Baseline
  Analysis will be primarily hypothesis generating and of a discovery nature. Gene expression will be compared to on-study vitamin D levels using Spearman correlation to look for associations between genes and Vitamin D. Gene expression will also be compared to polymorphisms in VDR using logistic regression to look for associations of host-genetics in the VDR region and general gene function in tumor.
Immune effector cell levels | Up to 36 months
  On-study regulatory T cells (Treg) and monocyte levels will be compared between sufficient and insufficient patients using Wilcoxon rank sum tests for each subtype. The pre and post-replacement levels will be assessed in CLL patients receiving replacement to look for a reduction in Tregs and monocytes, using a one-sample t-test on the difference testing for a mean of zero.
Serum cytokine profile | Up to 36 months
  A five-parameter regression formula will be used to calculate the sample concentrations from the standard curves and a change of 50% from the baseline value will be considered significant. Changes in all 30 cytokines in the kit will be evaluated with a focus on the tumor specific cytokines. In patients with abnormal cytokines, the pre and post-replacement cytokine level will be compared in patients receiving replacement to similar timepoints in patients not receiving replacement. The change in cytokine levels (post-pre) will be evaluated between the two groups using Wilcoxon rank sum tests.
Vitamin D metabolism single nucleotide polymorphisms (SNPs) | Up to 36 months
  All analyses will be performed separately for each lymphoma subtype. Individual vitamin D receptor (VDR) SNPs will be evaluated using a co-dominant model. Principal components will be used to generate a gene level assessment of VDR variability. Host genetic VDR markers will be compared to onstudy vitamin D levels to look for association between VDR polymorphisms and vitamin D stores using logistic regression. Host genetic VDR markers will be compared to outcome (time to first treatment [TFT], EFS, OS) using Cox regression models.
Vitamin D receptor expression on tumor cells | Baseline
  The results will be expressed as present or absent. In the case of immunohistochemistry for DLBCL, expression may be graded as 0-3+. In the case of CLL, the % cells positive will be reported. VDR expression from the tumor will be reported using summary tables. Expression will be compared with outcome (TFT, EFS, OS) using Cox models to examine if VDR expression is prognostic in these tumors. VDR expression will also be compared to polymorphisms in VDR using logistic regression or chi-square tests to look for associations of host-genetics in the VDR region and VDR function in tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E. Witzig, MD, Principal Investigator — Mayo Clinic
Locations (5):
- United States (5):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials